CLINICAL TRIAL: NCT00034567
Title: Alzheimer's Disease Prevention Instrument Protocol
Brief Title: Healthy Aging and Memory Study
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Other Study IDs: IA0032
Record Dates: First submitted 2002-04-30; First posted 2002-05-01 (Estimated); Last update posted 2007-09-18 (Estimated); Status verified 2007-09

CONDITIONS: Alzheimer Disease
Keywords: Prevention
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
This project will focus on the development and testing of efficient, cost effective measures that are specifically designed for use in Alzheimer's Disease (AD) primary prevention trials.

DETAILED DESCRIPTION:
This project will focus on the development and testing of efficient, cost effective measures that are specifically designed for use in AD primary prevention trials. The new or improved measures that have been developed will then be evaluated in 650 nondemented subjects enrolled in a simulated Alzheimer's disease prevention trial. Once enrolled, subjects will be followed for four years with annual clinical evaluations and interim six-month phone calls.

ELIGIBILITY:
Inclusion Criteria:

* 75 years or older.
* Fluent in English or Spanish.
* Stable medical condition for four weeks prior to screening visit.
* Stable medications for four weeks prior to screening visit.
* Either cognitively normal, or mild cognitive impairment. If MCI, the subject's CDR at screening have a global score of 0.5.
* mMMSE score greater than 88 for subjects with at least 8 years education, or greater than 80 for subjects with less than 8 years education, and FCSRT total free plus cued recall score greater than 44 with 3 learning trials.
* Willing to participate in four to five year follow-up study.
* Willing to identify person who can serve as informant.
* At least six years education or work history sufficient to exclude mental retardation

Exclusion Criteria:

* Meets DSM IV criteria for dementia
* History of clinically significant medical illness that would interfere with participation in trial, including active malignancy, myocardial infarction, or cerebrovascular accident within the past year
* Alcohol or substance abuse and/or active major psychiatric disorders
* Concurrent participation in a clinical drug trial
* History of mental retardation

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 650

CONTACTS AND LOCATIONS:
Overall Officials: Steven H. Ferris, PhD, Study Director — NYU Langone Health
Locations (39):
- United States (39):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Sun Health Research Institute, Sun City, Arizona
  - University of California, Irvine, Irvine, California
  - University of California, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Stanford/Va Aging Clinical Research Center, Palo Alto, California
  - University of California, Davis, Sacramento, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Baumel-Eisner Neuromedical Institute, Boca Raton, Boca Raton, Florida
  - Baumel-Eisner Ft Lauderdale, Fort Lauderdale, Florida
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Wien Center for Memory Disorders, Miami Beach, Florida
  - Baumel-Eisner Neuromedical Institute, Miami Beach, Miami Beach, Florida
  - University of South Florida, Tampa, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush Alzheimer's Disease Center, Chicago, Illinois
  - Indiana University Alzheimer's Center, Indianapolis, Indiana
  - University of Kentucky, Lexington, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Michigan Alzheimer's Disease Research Center, Ann Arbor, Michigan
  - Mayo Alzheimer's Disease Center, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nevada, Las Vegas, Las Vegas, Nevada
  - New York University School of Medicine, New York, New York
  - Mt. Sinai Medical Center, New York, New York
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Memorial Hospital of Rhode Island (Brown University), Pawtucket, Rhode Island
  - Medical University of South Carolina, North Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Result] Ferris SH, Aisen PS, Cummings J, Galasko D, Salmon DP, Schneider L, Sano M, Whitehouse PJ, Edland S, Thal LJ; Alzheimer's Disease Cooperative Study Group. ADCS Prevention Instrument Project: overview and initial results. Alzheimer Dis Assoc Disord. 2006 Oct-Dec;20(4 Suppl 3):S109-23. doi: 10.1097/01.wad.0000213870.40300.21. PMID 17135805
- [Result] Schneider LS, Clark CM, Doody R, Ferris SH, Morris JC, Raman R, Reisberg B, Schmitt FA. ADCS Prevention Instrument Project: ADCS-clinicians' global impression of change scales (ADCS-CGIC), self-rated and study partner-rated versions. Alzheimer Dis Assoc Disord. 2006 Oct-Dec;20(4 Suppl 3):S124-38. doi: 10.1097/01.wad.0000213878.47924.44. PMID 17135806
- [Result] Galasko D, Bennett DA, Sano M, Marson D, Kaye J, Edland SD; Alzheimer's Disease Cooperative Study. ADCS Prevention Instrument Project: assessment of instrumental activities of daily living for community-dwelling elderly individuals in dementia prevention clinical trials. Alzheimer Dis Assoc Disord. 2006 Oct-Dec;20(4 Suppl 3):S152-69. doi: 10.1097/01.wad.0000213873.25053.2b. PMID 17135809
- [Result] Sano M, Zhu CW, Whitehouse PJ, Edland S, Jin S, Ernstrom K, Thomas RG, Thal LJ, Ferris SH; Alzheimer Disease Cooperative Study Group. ADCS Prevention Instrument Project: pharmacoeconomics: assessing health-related resource use among healthy elderly. Alzheimer Dis Assoc Disord. 2006 Oct-Dec;20(4 Suppl 3):S191-202. doi: 10.1097/01.wad.0000213875.63171.87. PMID 17135812
- [Result] Walsh SP, Raman R, Jones KB, Aisen PS; Alzheimer's Disease Cooperative Study Group. ADCS Prevention Instrument Project: the Mail-In Cognitive Function Screening Instrument (MCFSI). Alzheimer Dis Assoc Disord. 2006 Oct-Dec;20(4 Suppl 3):S170-8. doi: 10.1097/01.wad.0000213879.55547.57. PMID 17135810
- [Result] Cummings JL, Raman R, Ernstrom K, Salmon D, Ferris SH; Alzheimer's Disease Cooperative Study Group. ADCS Prevention Instrument Project: behavioral measures in primary prevention trials. Alzheimer Dis Assoc Disord. 2006 Oct-Dec;20(4 Suppl 3):S147-51. doi: 10.1097/01.wad.0000213872.17429.0f. PMID 17135808
- [Result] Patterson MB, Whitehouse PJ, Edland SD, Sami SA, Sano M, Smyth K, Weiner MF; Alzheimer's Disease Cooperative Study Group. ADCS Prevention Instrument Project: quality of life assessment (QOL). Alzheimer Dis Assoc Disord. 2006 Oct-Dec;20(4 Suppl 3):S179-90. doi: 10.1097/01.wad.0000213874.25053.e5. PMID 17135811
- See also: UCSD Alzheimer's Disease Cooperative Study — http://adcs.ucsd.edu